CLINICAL TRIAL: NCT01059591
Title: A Single Blind, Randomised, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK424887 in Healthy Male Subjects and an Open Label Positron Emission Tomography Study to Evaluate the Serotonin Transporter and Neurokinin- Receceptor Occupancy
Brief Title: First Study in Humans With GSK424887
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 105011
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: NK1 antagonist and SSRI; Healthy subjects; Safety; First time in Human
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — N-(1-(3-chloro-1-naphthalenyl)ethyl)-2-(4-(4-fluorophenyl)-1-methyl-4-piperidinyl)-N-methylacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): GSK424887 once daily
  Interventions: Drug: GSK424887; Radiation: PET
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK424887 — GSK424887 2mg, 10mg, 50mg, 100mg capsule
  Arms: Active
Drug: Placebo — Placebo to match GSK424887 2mg, 10mg,50mg, 100mg capsule
  Arms: Placebo
Radiation: PET — Each subject will undergo 3 PET scans : one at Baseline and the others following dosing with GSK424887 at approximately 2h post-dose and aproximately 24 hours post-dose
  Arms: Active

SUMMARY:
This is the first study in Humans with GSK424887 to evaluate what effects, good or bad, the drug has on human health (safety and tolerability) and the amount of drug which gets into the bloodstream and is eliminated from the body (pharmacokinetics). Also the study aims to investigate the penetration of the drug in the human brain by using PET (Positron Emission Tomography) imaging technology

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-45 years, limited to 25-40 years for PET section

Exclusion Criteria:

* The subject has a positive: drug/alcohol, Hepatitis, HIV screen
* The subject has a history of psychiatric illness suicidal attempts or behaviour.
* Abuse of alcohol.
* Clinically significant laboratory, ECG abnormality;
* The subject has recently received an investigational.
* Use of prescription or non-prescription drugs,
* History or presence of allergy to the study drug or drugs of this class,.
* Donation of more than 500 mL blood within the 90 days before dosing.
* An unwillingness of male subjects to comply with contraceptive requirements
* Average daily caffeine intake exceeding Protocol requirements.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-05-25 (Actual); Primary Completion 2007-01-25 (Actual); Study Completion 2007-01-25 (Actual)

PRIMARY OUTCOMES:
Adverse event monitoring, vital signs (blood pressure, heart rate, ECGs, clinical laboratory assessments (standard laboratory parameters); Area under the concentration-time curve (AUC), Maximum observed concentration (Cmax) , tmax | 12 weeks

SECONDARY OUTCOMES:
Brain receptor occupancy | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 105011 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/105011?search=study&search_terms=105011#rs